CLINICAL TRIAL: NCT04338672
Title: The Impact of the Coronavirus Disease 2019 (Covid-19) Outbreak on Emergency Room Attendances of Surgical Patients at a Tertiary Medical Center
Brief Title: The Impact of the Covid-19 Outbreak on Emergency Room Attendances of Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SMC-20-7078-YZ-CTIL
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Emergency Service, Hospital; General Surgery
Keywords: Emergency; Surgery; Covid-19
MeSH Terms: conditions — Emergencies; COVID-19 | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pandemic Period: Patients who presented to the emergency department at our medical institute Sheba Medical Center between January 1 - March 31 in 2020.
  Interventions: Other: COVID-19 Pandemic
- Pre Pandemic Period: Patients who presented to the emergency department at our medical institute Sheba Medical Center between January 1 - March 31 in the following years: 2017, 2018, 2019,

INTERVENTIONS:
Other: COVID-19 Pandemic — Exposure: the novel coronavirus disease (Covid-19) outbreak
  Groups: Pandemic Period

SUMMARY:
Since December 2019, when the novel coronavirus disease (Covid-19) spread throughout the world, data have been needed on the effects of the pandemic on various aspects of healthcare systems. Recommendations for social distancing and quarantine decrees made by local governments, alongside the general public fear from the spread of the virus, are presumed to have markedly affected the trends in hospitals visits. Understanding the exact nature of the effect is critical for better anticipating and preparing health systems in the event of future outbreaks and in the post outbreak period. Therefore we intend to To identify retrospectively all patients who presented to the emergency department at our medical institute between January 1 - March 31 in the following years: 2017, 2018, 2019, 2020. We will examine the impact of COVID-19 on the rates of surgical emergency visits, ratio of surgical visits to non-surgical visits, the ratio of severe presentations to non-severe presentations, and the impact of age on ED attendance.

DETAILED DESCRIPTION:
Since December 2019, when the novel coronavirus disease (Covid-19) spread throughout the world, data have been needed on the effects of the pandemic on various aspects of healthcare systems. Recommendations for social distancing and quarantine decrees made by local governments, alongside the general public fear from the spread of the virus, are presumed to have markedly affected the trends in hospitals visits. Understanding the exact nature of the effect is critical for better anticipating and preparing health systems in the event of future outbreaks and in the post outbreak period. Additionally, deferring hospitals visits can potentially put patients at increased risk for morbidity and mortality, especially in postsurgical patients. Evaluating the impact of the pandemic on patient volume can guide decision-making in future scenarios.

Previous infectious disease outbreaks have been shown to impact ED volumes: The US Hantavirus outbreak in 1993 led to a 2-fold increase in ED visits; Escherichia coli 0157:H7 outbreak in Washington state in 1993 increased ED visits by 17%; However, the 2003 SARS outbreaks in Hong Kong, Taiwan, and Toronto reduced tertiary care ED visits by up to 47 percent.

ELIGIBILITY:
Inclusion Criteria:

* All patients visiting the ER of Sheba Medical Center between January 1 - March 31 in the following years: 2017, 2018, 2019, 2020

Exclusion Criteria:

* Patients less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged >18 years old who attended the emergency department of Sheba Medical Center between January 1 - March 31 in the following years: 2017, 2018, 2019, 2020
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-04-05 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Rates of emergency visits needing surgical consult | January 1 - March 31 in the following years: 2017, 2018, 2019, 2020
The ratio of severe presentations to non-severe presentations | January 1 - March 31 in the following years: 2017, 2018, 2019, 2020

SECONDARY OUTCOMES:
The impact of age on ED attendance rates | January 1 - March 31 in the following years: 2017, 2018, 2019, 2020
Differences in ED surgical visits (in terms of capacity and severity) of surgical patients depending on the presentation and the co morbidity | January 1 - March 31 in the following years: 2017, 2018, 2019, 2020

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heiber M, Lou WY. Effect of the SARS outbreak on visits to a community hospital emergency department. CJEM. 2006 Sep;8(5):323-8. doi: 10.1017/s148180350001397x. PMID 17338843
- [Background] Chen WK, Cheng YC, Chung YT, Lin CC. The impact of the SARS outbreak on an urban emergency department in Taiwan. Med Care. 2005 Feb;43(2):168-72. doi: 10.1097/00005650-200502000-00010. PMID 15655430
- [Derived] Anteby R, Zager Y, Barash Y, Nadler R, Cordoba M, Klang E, Klein Y, Ram E, Gutman M, Horesh N. The Impact of the Coronavirus Disease 2019 Outbreak on the Attendance of Patients with Surgical Complaints at a Tertiary Hospital Emergency Department. J Laparoendosc Adv Surg Tech A. 2020 Sep;30(9):1001-1007. doi: 10.1089/lap.2020.0465. Epub 2020 Jun 23. PMID 32589496